CLINICAL TRIAL: NCT02709655
Title: Interventional, Randomized, Double-blind, Placebo-controlled, Active-reference (Fluoxetine), Fixed-dose Study of Vortioxetine in Paediatric Patients Aged 7 to 11 Years, With Major Depressive Disorder (MDD)
Brief Title: Active Reference (Fluoxetine) Fixed-dose Study of Vortioxetine in Paediatric Participants Aged 7 to 11 Years With Major Depressive Disorder (MDD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12709A; 2008-005353-38 (EudraCT Number)
Record Dates: First submitted 2016-03-11; First posted 2016-03-16 (Estimated); Results first posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-08

CONDITIONS: Depressive Disorder, Major
Keywords: paediatric
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Vortioxetine; Fluoxetine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Vortioxetine 10 mg/day (Experimental)
  Interventions: Drug: Vortioxetine 10 mg/day
- Vortioxetine 20 mg/day (Experimental)
  Interventions: Drug: Vortioxetine 20 mg/day
- Fluoxetine 20 mg/day, (Active Comparator): A decision has been taken to stop recruitment into this treatment arm.
  Interventions: Drug: Fluoxetine 20mg/day
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Vortioxetine 10 mg/day — 10 mg/day, encapsulated tablet, orally (with addition of lower initial dose levels).
  Based on tolerability the dose may be reduced by 5 mg/day. No dose increase will be allowed
  Other Names: Brintellix ®; Lu AA21004
  Arms: Vortioxetine 10 mg/day
Drug: Vortioxetine 20 mg/day — 20 mg/day, encapsulated tablet, orally (with addition of lower initial dose levels).
  Based on tolerability the dose may be reduced by 5 mg/day. No dose increase will be allowed
  Other Names: Brintellix ®; Lu AA21004
  Arms: Vortioxetine 20 mg/day
Drug: Fluoxetine 20mg/day — 20 mg/day, encapsulated tablet, orally (with addition of lower initial dose levels).
  Based on tolerability the dose may be reduced by 10 mg/day. No dose increase will be allowed
  Arms: Fluoxetine 20 mg/day,
Other: Placebo — Encapsulated tablet, orally
  Arms: Placebo

SUMMARY:
Investigation of the efficacy and safety of a new potential treatment of Major depressive disorder (MDD) in paediatric participants (age 7 to 11 years).

ELIGIBILITY:
Inclusion Criteria:

1. The participant has MDD, diagnosed according to Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5™).
2. The participant has a CDRS-R total score ≥45 at the Screening Visit and the Baseline.
3. The participant has a CGI-S score ≥4 at the Screening Visit and the Baseline.
4. The participant is a boy or girl, aged ≥7 and <12 years at Screening Visit
5. The participant has provided assent to participation and parent(s)/legal representative (s) signed the Informed Consent Form.

Exclusion Criteria:

1. The participant has participated in a clinical study <30 days prior to the Screening Visit.
2. The participant has previously participated in a study with vortioxetine.

Other protocol defined inclusion and exclusion criteria may apply

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 683 (Actual)
Dates: Start 2016-05-18 (Actual); Primary Completion 2022-01-21 (Actual); Study Completion 2022-01-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (98):
- United States (34):
  - Woodland International Research Group, Little Rock, Arkansas
  - Sun Valley Research Center, Imperial, California
  - Synergy Clinical Research Center, Lemon Grove, California
  - Alliance for Wellness dba Alliance for Research, Long Beach, California
  - NRC Research Institute, Orange, California
  - Asclepes Research Center, Panorama City, California
  - Children's National Medical Center Merge, Washington D.C., District of Columbia
  - Sarkis Clinical Trials, Gainesville, Florida
  - Medical Research Group of Central Florida, Orange City, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Northwest Behavioral Research Center, Marietta, Georgia
  - American Medical Research, Inc., Chicago, Illinois
  - AMR- Baber Research, Inc., Naperville, Illinois
  - AMR Conventions Research, Warrenville, Illinois
  - Kansas University School of Medicine-Wichita, Wichita, Kansas
  - Lake Charles Clinical Trials, Lake Charles, Louisiana
  - Kennedy Krieger Institute, Baltimore, Maryland
  - St. Charles Psychiatric Associates - Midwest Research Group, Saint Charles, Missouri
  - Millennium Psychiatric Associates, LLC, St Louis, Missouri
  - Princeton Medical Institute, Princeton, New Jersey
  - Manhattan Behavioral Medicine, New York, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - University Hospital Cleveland Medical Center Division of Child and Adolescent Psychiatry, Cleveland, Ohio
  - North Star Medical Research, LLC, Middleburg Heights, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Paradigm Research Professionals, LLC, Oklahoma City, Oklahoma
  - Research Strategies Of Memphis, Llc, Memphis, Tennessee
  - BioBehavioral Research of Austin, Austin, Texas
  - AIM Trials, LLC, Plano, Texas
  - Research Across America, Plano, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Westside Medical, Clinton, Utah
  - Aspen Clinical Research, LLC, Orem, Utah
- Bulgaria (2):
  - MHAT Targovishte AD, Targovisthe
  - Diagnostic Consultative Center Mladost-M Varna OOD, Varna
- Paediatric Sleep Research Inc., Toronto, Ontario, Canada
- Colombia (4):
  - E.S.E. Hospital Mental de Antioquia HOMO, Bello, Antioquia
  - Centro de Investigaciones y Proyectos en Neurociencias CIPNA LTDA IPS., Barranquilla, Atlántico
  - Centro de investigaciones del Sistema Nervioso SAS Grupo CISNE SAS, Bogotá, DC
  - Psynapsis Salud Mental S.A., Pereira, Risaralda Department
- Marienthali Kliinik, Tallinn, Estonia
- France (3):
  - Cabinet Psyche, Douai, Nord
  - Centre Medical Ambroise Pare, Élancourt
  - CHU de Nantes - Hopital Hotel Dieu, Nantes
- Rheinhessen-Fachklinik Mainz, Kinder und Jugendpsychiatri, Mainz, Germany
- Hungary (2):
  - Vadaskert Alapitvany, Budapest
  - Bekes Megyei Kozponti Korhaz Pandy Kalman Tagkorhaza, Gyula
- Israel (3):
  - Shalvata Mental Health Center, Hod HaSharon
  - Ramat Chen - Mental Health Clinic, Tel Aviv
  - The Chaim Sheba Medical Center - The Edmond and Lily Safra Children's Hospital, Tel Litwinsky
- Italy (3):
  - Scientific Institute Fondazione Stella Maris, Calambrone Pisa, Pisa
  - Sciaf Ulss 16 Padova, Padua, Regione Veneto
  - University Federico II Of Naples, Napoli
- Latvia (2):
  - Linda Keruze's Psychiatric Center, LLC, Liepāja
  - Children Hospilal -Gailezers, Riga
- Mexico (9):
  - Centro Investigacion Medico Biologica Y Terapia Avanzada, Guadalajara, Jalisco
  - Clinica Cemelli, Guadalajara, Jalisco
  - Roberto Zepeda Sanchez, Guadalajara, Jalisco
  - Instituto Nacional de Pediatria (INP) (National Institute of Pediatrics), Mexico City, Mexico City
  - CRI Centro Regiomontano de Investigacion SC, Monterrey, Nuevo León
  - Centro para el Desarrollo de la Medicina y de Asistencia Medica Especializada S.C, Culiacan de Rosales, Sinaloa
  - B & B Investigaciones Medicas, SC, Mazatlán, Sinaloa
  - ICARO Investigaciones en Medicina S.A. de C.V., Chihuahua City
  - BIND Investigaciones S.C, San Luis Potosí City
- Poland (6):
  - Prywatne Gabinety Lekarskie Promedicus, Bialystok, Podlaskie Voivodeship
  - Centrum Badan Klinicznych PI-House Sp. z o.o., Gdansk
  - Przychodnia Syntonia Poradnia Zdrowia Psychicznego, Kielce
  - Spectrum Centrum Psychiatrii Specjalistyczny Gabinet Psychiatryczny, Lublin
  - Filip Rybakowski Specjalistyczna Praktyka Lekarska, Poznan
  - Specjalistyczny Szpital im. dra A. Sokolowskiego w Walbrzychu, Wałbrzych
- Russia (13):
  - Medicorehabilitation Research Center Phoenix, Rostov-on-Don, Rostov State
  - Stavropol Region Psychiatric Hospital No.2, Stavropol, Stavropol Kray
  - Arkhangelsk Regional Clinical Mental Hospital, Arkhangelsk
  - GUZ Engels Psychiatric Hospital, Engel's
  - State Budgetary Healthcare Institution (SBHI) Specialized Clinical Psychiatric Hospital 1 of the ..., Krasnodar
  - LLC City Neurological Center Sibneuromed, Novosibirsk
  - Rostov State Medical University of the Minzdravsotsrazvitiya of Russia, Rostov-on-Don
  - City Psychiatric Hospital No.3 named after I.I. Skvortsov-Stepanov, Saint Petersburg
  - Saratov State Medical University, Saratov
  - Guz Saratov Regional Psychiatric Hospital St. Sofii, Saratov
  - Nebbiolo LLC, Tomsk
  - Yaroslavl Regional Clinical Psychiatry Hospital, Yaroslavl
  - State Budgetary Healthcare Institution of Sverdlovsk Region Â¿Sverdlovsk Regional Clinical Psychi..., Yekaterinburg
- Serbia (5):
  - Child and Adolescent Neurology and Psychiatry Clinic, Belgrade
  - Institute of Mental Health, Belgrade
  - University Clinical Center Kragujevac, Kragujevac
  - Clinical Center of Vojvodina - Clinic of Psychiatry, Novi Sad
  - Daily Hospital for Children and Adolescents, Pantelej-Nis
- South Africa (2):
  - Cape Trial Centre, Bellville, Cape Town
  - Tara Hospital, Sandhurst, Gauteng
- Seoul National University Hospital, Seoul, South Korea
- Spain (2):
  - Hospital Universitario Fundacion Alcorcon, Alcorcón, Madrid
  - Unidad de Salud Mental Infanto-Juvenil (USMI-J) Edificio de Consultas Externas. Hospital MarAtimo, Torremolinos, Malaga
- Ukraine (4):
  - Ukrainian Research Institute Of Social, Forensic Psychiatry And Drug Abuse, Kiev City Psychoneuro..., Kyiv
  - Odessa Regional Medical Centre of Mental Health, Odesa
  - Maltsev Poltava Regional Clinical Psychiatric Hospital, Higher State Educational Institution Of U..., Poltava
  - Ternopil Regional Clinical Municipal Psycho-Neurological Hospital, Ternopil State Medical Univers..., Ternopil

REFERENCES:
- [Derived] Huss M, Findling RL, DelBello MP, Necking O, Petersen ML, Schmidt SN, Rosen M. Vortioxetine for Major Depressive Disorder in Children: 12-Week Randomized, Placebo-Controlled Study. JAACAP Open. 2024 Nov 22;3(3):736-748. doi: 10.1016/j.jaacop.2024.11.002. eCollection 2025 Sep. PMID 40922774

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study included 2 periods: single-blind (SB) (treatment with standardized brief psychosocial intervention [BPI] and placebo) and double-blind (DB) (treatment with BPI and placebo, vortioxetine 10 milligrams [mg]/day, vortioxetine 20 mg/day, or fluoxetine 20 mg/day).
Pre-assignment Details: Participants who demonstrated an incomplete improvement in depressive symptoms at the end of the SB period (Week 4) entered the DB period to receive BPI (2 sessions) and treatment as follows: Prior to the interim analysis, participants were randomized in a 1:1:1:1 ratio to placebo, vortioxetine 10 mg/day, vortioxetine 20 mg/day, or fluoxetine 20 mg/day. After interim analysis, participants were randomized in a 1:1:1 ratio to placebo, vortioxetine 10 mg/day, or vortioxetine 20 mg/day.
Groups:
- Single-Blind: Placebo: Participants received BPI (3 sessions) and placebo capsules orally once daily for 4 weeks.
- Double-Blind: Placebo: Participants received placebo capsules orally once daily for 8 weeks. Participants received 2 sessions of BPI also.
- Double-Blind: Vortioxetine 10 mg: Participants initiated treatment with vortioxetine capsules 5 mg/day orally for 2 days and thereafter they received 10 mg/day for up to Week 8. Based on the tolerability, vortioxetine dose could be reduced by 5 mg/day at Week 4. Participants received 2 sessions of BPI also.
- Double-Blind: Vortioxetine 20 mg: Participants initiated treatment with vortioxetine capsules 5 mg/day orally for 2 days followed by 10 mg/day for 2 days and 15 mg/day for 2 days, and thereafter they received vortioxetine 20 mg/day for up to Week 8. Based on the tolerability, vortioxetine dose could be reduced by 5 mg/day at Week 4. Participants received 2 sessions of BPI also.
- Double-Blind: Fluoxetine 20 mg: Participants initiated treatment with fluoxetine 10 mg/day orally for 6 days and thereafter they received 20 mg/day. for up to Week 8. Based on the tolerability, fluoxetine dose could be reduced by 10 mg/day at Week 4. Participants received 2 sessions of BPI also.
Period: Single-Blind Phase (4 Weeks)
Arm/Group | Single-Blind: Placebo | Double-Blind: Placebo | Double-Blind: Vortioxetine 10 mg | Double-Blind: Vortioxetine 20 mg | Double-Blind: Fluoxetine 20 mg
Started | 683 | 0 | 0 | 0 | 0
Received at Least 1 Dose of Study Drug | 677 | 0 | 0 | 0 | 0
Completed | 540 | 0 | 0 | 0 | 0
Not Completed | 143 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 8 | 0 | 0 | 0 | 0
Not completed — Non-compliance with study drug | 3 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 3 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 15 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0
Not completed — Failure to meet randomization criteria | 85 | 0 | 0 | 0 | 0
Not completed — Other than specified | 20 | 0 | 0 | 0 | 0
Not completed — Enrolled but not treated | 6 | 0 | 0 | 0 | 0
Period: Double-Blind Phase (8 Weeks)
Arm/Group | Single-Blind: Placebo | Double-Blind: Placebo | Double-Blind: Vortioxetine 10 mg | Double-Blind: Vortioxetine 20 mg | Double-Blind: Fluoxetine 20 mg
Started | 0 | 153 | 151 | 153 | 83
Received at Least 1 Dose of Study Drug | 0 | 153 | 151 | 153 | 83
Full Analysis Set (FAS) (All participants randomized to the double-blind, 8-week treatment period (Phase B) who took at least 1 dose of double-blind study drug and who had a valid baseline (Week 4 of Phase A) assessment and at least 1 valid post-baseline assessment of the Children Depression Rating Scale - Revised (CDRS-R) total score) | 0 | 153 | 148 | 148 | 81
Completed | 0 | 138 | 135 | 133 | 78
Not Completed | 0 | 15 | 16 | 20 | 5
Not completed — Adverse Event | 0 | 1 | 2 | 3 | 0
Not completed — Lack of Efficacy | 0 | 2 | 0 | 0 | 1
Not completed — Non-compliance with study drug | 0 | 1 | 3 | 6 | 1
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 4 | 4 | 4 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 2 | 0
Not completed — Other than specified | 0 | 5 | 7 | 5 | 2

BASELINE CHARACTERISTICS:
Population: All-patients-treated set Phase A (APTS_A) included all participants enrolled to the 4-week Single-blind period (Phase A) who received at least 1 dose of study drug.
Arm/Group | Single-Blind: Placebo
Number analyzed (Participants) | 677
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.3 (1.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 312
  Male | 365
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 1
  Race: Asian | 2
  Race: Black or African American | 112
  Race: Not Reported | 12
  Race: Other | 229
  Race: White | 321
Children Depression Rating Scale - Revised (CDRS-R) Total Score [Mean (Standard Deviation); unit: units on a scale] — The CDRS-R was rated by a clinician following interviews with the child and parent and consisted of 17 items out of which 3 items rated nonverbal observations (listless speech, hypoactivity, and depressed affect). Fourteen items were rated on a 7-point scale from 1 to 7, and 3 items (sleep disturbance, appetite disturbance, and listless speech) were scored on a 5-point scale from 1 to 5. A rating of 1 indicated normal functioning and a higher number indicated a greater degree of depression. The total score ranged from 17 (normal) to 113 (severe depression). Population: Baseline measure was taken for all participants randomized to Phase B.
  units on a scale
    number analyzed (Participants) | 530
    (all) | 63.4 (9.12)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Children Depression Rating Scale - Revised (CDRS-R) Total Score at Week 8 of Phase B
Description: The CDRS-R is a clinician-rated scale to measure the severity of depression in children and adolescents. The CDRS-R was rated by a clinician following interviews with the child and parent and consisted of 17 items out of which 3 items rated nonverbal observations (listless speech, hypoactivity, and depressed affect). Fourteen items were rated on a 7-point scale from 1 to 7, and 3 items (sleep disturbance, appetite disturbance, and listless speech) were scored on a 5-point scale from 1 to 5. A rating of 1 indicated normal functioning and a higher number indicated a greater degree of depression. The total score ranged from 17 (normal) to 113 (severe depression). Least square (LS) mean was estimated using a restricted maximum likelihood (REML)-based Mixed Model Repeated Measurements (MMRM) approach.
Time Frame: Baseline (Week 4 of Phase A), Week 8 of Phase B
Population: Full analysis set (FAS) included all participants randomized to the double-blind, 8-week treatment period (Phase B) who took at least 1 dose of double-blind study drug and who had a valid baseline (Week 4 of Phase A) assessment and at least 1 valid post-baseline assessment of the CDRS-R total score. Overall number of participants analyzed = participants evaluated for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Vortioxetine Average (Avg. VOR): Avg. VOR is the average dose effect of the 2 vortioxetine doses (Vortioxetine 10 mg and Vortioxetine 20 mg).
Arm/Group | Double-Blind: Placebo | Double-Blind: Vortioxetine 10 mg | Double-Blind: Vortioxetine 20 mg | Double-Blind: Fluoxetine 20 mg | Vortioxetine Average (Avg. VOR)
Number analyzed (Participants) | 136 | 132 | 134 | 78 | 266
units on a scale | -17.48 (1.35) | -19.20 (1.37) | -19.94 (1.37) | -20.78 (1.60) | -19.57 (1.16)
Statistical Analysis 1: Comparison: Double-Blind: Placebo vs Vortioxetine Average (Avg. VOR); Analysis was performed using an REML-based MMRM approach with freely varying mean and covariance structure and with country, treatment (vortioxetine 10 mg/day, vortioxetine 20 mg/day, fluoxetine, and placebo), and Week as fixed factors and Baseline CDRS-R total score as a continuous covariate, the treatment-by-week interaction, and Baseline CDRS-R-by-Week interaction; Test type: Other; p = 0.0937, Mixed Models Analysis; Mean Difference (Final Values) = -2.09, 95% CI 2-sided [-4.54 to 0.36], Standard Error of Mean 1.24
Statistical Analysis 2: Comparison: Double-Blind: Placebo vs Double-Blind: Vortioxetine 10 mg; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.2336, Mixed Models Analysis; Mean Difference (Final Values) = -1.72, 95% CI 2-sided [-4.56 to 1.11], Standard Error of Mean 1.44
Statistical Analysis 3: Comparison: Double-Blind: Placebo vs Double-Blind: Vortioxetine 20 mg; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0879, Mixed Models Analysis; Mean Difference (Final Values) = -2.46, 95% CI 2-sided [-5.29 to 0.37], Standard Error of Mean 1.44
Statistical Analysis 4: Comparison: Double-Blind: Placebo vs Double-Blind: Fluoxetine 20 mg; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0531, Mixed Models Analysis; Mean Difference (Final Values) = -3.30, 95% CI 2-sided [-6.65 to 0.04], Standard Error of Mean 1.70

2. Secondary Outcome: Change From Baseline in CDRS-R Total Score at Weeks 2, 4, and 6 of Phase B
Description: The CDRS-R is a clinician-rated scale to measure the severity of depression in children and adolescents. The CDRS-R was rated by a clinician following interviews with the child and parent and consisted of 17 items out of which 3 items rated nonverbal observations (listless speech, hypoactivity, and depressed affect). Fourteen items were rated on a 7-point scale from 1 to 7, and 3 items (sleep disturbance, appetite disturbance, and listless speech) were scored on a 5-point scale from 1 to 5. A rating of 1 indicated normal functioning and a higher number indicated a greater degree of depression. The total score ranged from 17 (normal) to 113 (severe depression).
Time Frame: Baseline (Week 4 of Phase A), Weeks 2, 4, and 6 of Phase B
Population: FAS included all participants randomized to the double-blind, 8-week treatment period (Phase B) who took at least 1 dose of double-blind study drug and who had a valid baseline (Week 4 of Phase A) assessment and at least 1 valid post-baseline assessment of the CDRS-R total score. Overall number of participants analyzed = participants evaluated for this outcome measure. Number analyzed = participants evaluable at specified timepoint.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-Blind: Placebo | Double-Blind: Vortioxetine 10 mg | Double-Blind: Vortioxetine 20 mg | Double-Blind: Fluoxetine 20 mg
Number analyzed (Participants) | 153 | 147 | 146 | 80
units on a scale
  Change at Week 2 | -9.20 (1.17) | -9.54 (1.18) | -10.30 (1.19) | -10.17 (1.32)
  Change at Week 4: number analyzed (Participants) | 145 | 137 | 139 | 78
  Change at Week 4 | -13.15 (1.28) | -14.56 (1.30) | -15.62 (1.30) | -13.97 (1.50)
  Change at Week 6: number analyzed (Participants) | 143 | 136 | 137 | 78
  Change at Week 6 | -16.00 (1.32) | -17.64 (1.34) | -18.28 (1.34) | -17.75 (1.56)

3. Secondary Outcome: Change From Baseline in CDRS-R Subscores (Mood, Somatic, Subjective, and Behaviour) at Weeks 2, 4, 6, and 8 of Phase B
Description: The CDRS-R was rated by a clinician following interviews with the child and parent and consisted of 17 items out of which 3 items rated nonverbal observations (listless speech, hypoactivity, and depressed affect). Fourteen items were rated on a 7-point scale from 1 to 7, and 3 items (sleep disturbance, appetite disturbance, and listless speech) were scored on a 5-point scale from 1 to 5. A rating of 1 indicated normal functioning and a higher number indicated a greater degree of depression. The total score ranged from 17 (normal) to 113 (severe depression). Four subscores were defined based on the CDRS-R: Mood: sum of items 8, 11, 14, 15; score range 4 to 28, Somatic: sum of items 4, 5, 6, 7, 16, 17; score range 6 to 36, Subjective: sum of items 9, 10, 12, 13; score range 4 to 28, and Behaviour: sum of items 1, 2, 3; score range 3 to 21. Higher scores indicated the most severe measure of depression.
Time Frame: Baseline (Week 4 of Phase A), Weeks 2, 4, 6, and 8 of Phase B
Population: FAS included all participants randomized to the double-blind, 8-week treatment period (Phase B) who took at least 1 dose of double-blind study drug and who had a valid baseline (Week 4 of Phase A) assessment and at least 1 valid post-baseline assessment of the CDRS-R total score. Overall number of participants analyzed = participants evaluated for this outcome measure. Number analyzed = participants evaluable for specified categories.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-Blind: Placebo | Double-Blind: Vortioxetine 10 mg | Double-Blind: Vortioxetine 20 mg | Double-Blind: Fluoxetine 20 mg
Number analyzed (Participants) | 153 | 147 | 146 | 80
units on a scale
  Mood Score: Change at Week 2 | -2.82 (0.40) | -3.10 (0.40) | -3.47 (0.40) | -3.02 (0.45)
  Mood Score: Change at Week 4: number analyzed (Participants) | 145 | 137 | 139 | 78
  Mood Score: Change at Week 4 | -3.69 (0.42) | -4.39 (0.43) | -4.77 (0.43) | -3.73 (0.49)
  Mood Score: Change at Week 6: number analyzed (Participants) | 143 | 136 | 137 | 78
  Mood Score: Change at Week 6 | -4.67 (0.43) | -5.39 (0.44) | -5.52 (0.44) | -4.97 (0.51)
  Mood Score: Change at Week 8: number analyzed (Participants) | 136 | 132 | 134 | 78
  Mood Score: Change at Week 8 | -5.08 (0.44) | -5.64 (0.44) | -5.95 (0.45) | -5.84 (0.51)
  Somatic Score: Change at Week 2 | -2.81 (0.44) | -2.61 (0.44) | -2.88 (0.44) | -3.02 (0.50)
  Somatic Score: Change at Week 4: number analyzed (Participants) | 145 | 137 | 139 | 78
  Somatic Score: Change at Week 4 | -4.08 (0.47) | -4.30 (0.48) | -4.70 (0.48) | -4.26 (0.56)
  Somatic Score: Change at Week 6: number analyzed (Participants) | 143 | 136 | 137 | 78
  Somatic Score: Change at Week 6 | -4.86 (0.48) | -5.53 (0.49) | -5.33 (0.49) | -5.57 (0.57)
  Somatic Score: Change at Week 8: number analyzed (Participants) | 136 | 132 | 134 | 78
  Somatic Score: Change at Week 8 | -5.38 (0.49) | -6.15 (0.50) | -6.08 (0.50) | -6.44 (0.57)
  Subjective Score: Change at Week 2 | -1.44 (0.22) | -1.46 (0.22) | -1.43 (0.22) | -1.56 (0.25)
  Subjective Score: Change at Week 4: number analyzed (Participants) | 145 | 137 | 139 | 78
  Subjective Score: Change at Week 4 | -2.04 (0.23) | -2.12 (0.23) | -2.20 (0.23) | -2.17 (0.27)
  Subjective Score: Change at Week 6: number analyzed (Participants) | 143 | 136 | 137 | 78
  Subjective Score: Change at Week 6 | -2.43 (0.24) | -2.42 (0.24) | -2.65 (0.24) | -2.38 (0.28)
  Subjective Score: Change at Week 8: number analyzed (Participants) | 136 | 132 | 134 | 78
  Subjective Score: Change at Week 8 | -2.56 (0.24) | -2.59 (0.24) | -2.84 (0.24) | -2.65 (0.28)
  Behaviour Score: Change at Week 2 | -2.16 (0.34) | -2.40 (0.34) | -2.56 (0.35) | -2.61 (0.39)
  Behaviour Score: Change at Week 4: number analyzed (Participants) | 145 | 137 | 139 | 78
  Behaviour Score: Change at Week 4 | -3.39 (0.38) | -3.77 (0.39) | -4.00 (0.39) | -3.80 (0.45)
  Behaviour Score: Change at Week 6: number analyzed (Participants) | 143 | 136 | 137 | 78
  Behaviour Score: Change at Week 6 | -4.09 (0.39) | -4.31 (0.39) | -4.83 (0.40) | -4.80 (0.46)
  Behaviour Score: Change at Week 8: number analyzed (Participants) | 136 | 132 | 134 | 78
  Behaviour Score: Change at Week 8 | -4.47 (0.40) | -4.80 (0.41) | -5.09 (0.41) | -5.83 (0.48)

4. Secondary Outcome: Percentage of Participants With CDRS-R Response
Description: CDRS-R response was defined as a ≥50% decrease in CDRS-R total score, calculated as: (change from baseline [Randomization])/(baseline value - 17). The CDRS-R is a clinician-rated scale to measure the severity of depression in children and adolescents. The CDRS-R was rated by a clinician following interviews with the child and parent and consisted of 17 items out of which 3 items rated nonverbal observations (listless speech, hypoactivity, and depressed affect). Fourteen items were rated on a 7-point scale from 1 to 7, and 3 items (sleep disturbance, appetite disturbance, and listless speech) were scored on a 5-point scale from 1 to 5. A rating of 1 indicated normal functioning and a higher number indicated a greater degree of depression. The total score ranged from 17 (normal) to 113 (severe depression).
Time Frame: Weeks 2, 4, 6, and 8 of Phase B
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind: Placebo | Double-Blind: Vortioxetine 10 mg | Double-Blind: Vortioxetine 20 mg | Double-Blind: Fluoxetine 20 mg
Number analyzed (Participants) | 153 | 147 | 146 | 80
percentage of participants
  Week 2 | 7.8 | 10.2 | 11.6 | 16.3
  Week 4: number analyzed (Participants) | 145 | 137 | 139 | 78
  Week 4 | 20.7 | 23.4 | 26.6 | 26.9
  Week 6: number analyzed (Participants) | 143 | 136 | 137 | 78
  Week 6 | 30.8 | 31.6 | 37.2 | 33.3
  Week 8: number analyzed (Participants) | 136 | 132 | 134 | 78
  Week 8 | 29.4 | 36.4 | 41.0 | 47.4

5. Secondary Outcome: Percentage of Participants With CDRS-R Remission
Description: CDRS-R remission was defined as a CDRS-R total score ≤28. The CDRS-R is a clinician-rated scale to measure the severity of depression in children and adolescents. The CDRS-R was rated by a clinician following interviews with the child and parent and consisted of 17 items out of which 3 items rated nonverbal observations (listless speech, hypoactivity, and depressed affect). Fourteen items were rated on a 7-point scale from 1 to 7, and 3 items (sleep disturbance, appetite disturbance, and listless speech) were scored on a 5-point scale from 1 to 5. A rating of 1 indicated normal functioning and a higher number indicated a greater degree of depression. The total score ranged from 17 (normal) to 113 (severe depression).
Time Frame: Weeks 2, 4, 6, and 8 of Phase B
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind: Placebo | Double-Blind: Vortioxetine 10 mg | Double-Blind: Vortioxetine 20 mg | Double-Blind: Fluoxetine 20 mg
Number analyzed (Participants) | 153 | 147 | 146 | 80
percentage of participants
  Week 2 | 2.0 | 5.4 | 2.7 | 3.8
  Week 4: number analyzed (Participants) | 145 | 137 | 139 | 78
  Week 4 | 9.0 | 9.5 | 10.1 | 9.0
  Week 6: number analyzed (Participants) | 143 | 136 | 137 | 78
  Week 6 | 14.7 | 15.4 | 15.3 | 14.1
  Week 8: number analyzed (Participants) | 136 | 132 | 134 | 78
  Week 8 | 14.7 | 16.7 | 20.1 | 26.9

6. Secondary Outcome: Change From Baseline in General Behaviour Inventory (GBI) Depression Subscale Score, Using the 10-Item Depression Subscale Assessed by Parent (PGBI-10D) and Child (CGBI-10D) at Weeks 2, 4, 6, and 8 of Phase B
Description: The GBI 10-item depression scale was developed to screen for depressive symptoms in children and adolescents. Two versions of the GBI 10-item depression scale were used, the child rated version (CGBI) and the parent rated version (PGBI). The 10 depression items were rated on a 4-point scale from 0 (never or hardly ever) to 3 (very often or almost constantly). The total score ranged from 0 to 30, with higher scores indicating greater pathology.
Time Frame: Baseline (Week 4 of Phase A), Weeks 2, 4, 6, and 8 of Phase B
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-Blind: Placebo | Double-Blind: Vortioxetine 10 mg | Double-Blind: Vortioxetine 20 mg | Double-Blind: Fluoxetine 20 mg
Number analyzed (Participants) | 152 | 147 | 146 | 80
units on a scale
  PGBI: Change at Week 2 | -3.33 (0.55) | -3.38 (0.55) | -3.78 (0.56) | -3.78 (0.63)
  PGBI: Change at Week 4: number analyzed (Participants) | 143 | 137 | 137 | 78
  PGBI: Change at Week 4 | -4.11 (0.58) | -4.72 (0.59) | -5.33 (0.59) | -4.45 (0.68)
  PGBI: Change at Week 6: number analyzed (Participants) | 142 | 136 | 137 | 78
  PGBI: Change at Week 6 | -5.32 (0.58) | -5.58 (0.59) | -5.82 (0.59) | -6.05 (0.68)
  PGBI: Change at Week 8: number analyzed (Participants) | 136 | 132 | 134 | 78
  PGBI: Change at Week 8 | -5.81 (0.61) | -6.51 (0.62) | -6.46 (0.62) | -6.56 (0.72)
  CGBI: Change at Week 2: number analyzed (Participants) | 149 | 145 | 143 | 76
  CGBI: Change at Week 2 | -2.66 (0.61) | -3.32 (0.61) | -3.27 (0.61) | -2.94 (0.70)
  CGBI: Change at Week 4: number analyzed (Participants) | 141 | 136 | 134 | 75
  CGBI: Change at Week 4 | -3.65 (0.65) | -4.15 (0.65) | -4.16 (0.65) | -3.16 (0.76)
  CGBI: Change at Week 6: number analyzed (Participants) | 139 | 134 | 135 | 75
  CGBI: Change at Week 6 | -4.62 (0.63) | -5.43 (0.64) | -5.17 (0.63) | -5.14 (0.73)
  CGBI: Change at Week 8: number analyzed (Participants) | 134 | 131 | 132 | 75
  CGBI: Change at Week 8 | -5.26 (0.65) | -6.12 (0.66) | -5.48 (0.65) | -5.46 (0.76)

7. Secondary Outcome: Parent Global Assessment (PGA) Score
Description: The PGA is a parent-rated variation of the CGI-I to evaluate the severity of the child's symptoms. The PGA reflects assessments of symptoms using a 7-point scale ranging from 1 (very much improved) to 7 (very much worse).
Time Frame: Weeks 2, 4, 6, and 8 of Phase B
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-Blind: Placebo | Double-Blind: Vortioxetine 10 mg | Double-Blind: Vortioxetine 20 mg | Double-Blind: Fluoxetine 20 mg
Number analyzed (Participants) | 152 | 147 | 145 | 80
units on a scale
  Week 2 | 3.31 (0.09) | 3.25 (0.09) | 3.18 (0.09) | 3.13 (0.11)
  Week 4: number analyzed (Participants) | 143 | 137 | 136 | 78
  Week 4 | 2.97 (0.10) | 2.90 (0.10) | 2.84 (0.10) | 2.90 (0.12)
  Week 6: number analyzed (Participants) | 142 | 136 | 136 | 78
  Week 6 | 2.73 (0.10) | 2.73 (0.10) | 2.68 (0.10) | 2.80 (0.12)
  Week 8: number analyzed (Participants) | 136 | 132 | 133 | 78
  Week 8 | 2.68 (0.11) | 2.62 (0.11) | 2.61 (0.11) | 2.59 (0.13)

8. Secondary Outcome: Change From Baseline in Clinical Global Impression - Severity of Illness (CGI-S) Score at Weeks 1, 2, 3, 4, 6, and 8 of Phase B
Description: The CGI-S provides the clinician's impression of the participant's current state of mental illness. The clinician uses his or her clinical experience of this participant population to rate the severity of the participant's current mental illness on a 7-point scale ranging from 1 (normal - not at all ill) to 7 (among the most extremely ill participants).
Time Frame: Baseline (Week 4 of Phase A), Weeks 1, 2, 3, 4, 6, and 8 of Phase B
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-Blind: Placebo | Double-Blind: Vortioxetine 10 mg | Double-Blind: Vortioxetine 20 mg | Double-Blind: Fluoxetine 20 mg
Number analyzed (Participants) | 153 | 148 | 146 | 81
units on a scale
  Change at Week 1 | -0.25 (0.07) | -0.27 (0.07) | -0.28 (0.07) | -0.22 (0.08)
  Change at Week 2: number analyzed (Participants) | 153 | 146 | 144 | 81
  Change at Week 2 | -0.50 (0.08) | -0.60 (0.08) | -0.65 (0.08) | -0.63 (0.10)
  Change at Week 3: number analyzed (Participants) | 150 | 145 | 145 | 78
  Change at Week 3 | -0.67 (0.08) | -0.62 (0.08) | -0.79 (0.08) | -0.77 (0.10)
  Change at Week 4: number analyzed (Participants) | 145 | 137 | 139 | 78
  Change at Week 4 | -0.95 (0.09) | -1.00 (0.09) | -1.06 (0.09) | -1.01 (0.12)
  Change at Week 6: number analyzed (Participants) | 143 | 136 | 137 | 78
  Change at Week 6 | -1.13 (0.10) | -1.22 (0.10) | -1.27 (0.10) | -1.23 (0.12)
  Change at Week 8: number analyzed (Participants) | 137 | 132 | 134 | 78
  Change at Week 8 | -1.31 (0.10) | -1.40 (0.11) | -1.44 (0.11) | -1.57 (0.13)

9. Secondary Outcome: Clinical Global Impression - Global Improvement (CGI-I) Score
Description: The CGI-I provides the clinician's impression of the participant's improvement (or worsening). The clinician assesses the participant's condition relative to a baseline on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse).
Time Frame: Weeks 1, 2, 3, 4, 6, and 8 of Phase B
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-Blind: Placebo | Double-Blind: Vortioxetine 10 mg | Double-Blind: Vortioxetine 20 mg | Double-Blind: Fluoxetine 20 mg
Number analyzed (Participants) | 153 | 148 | 145 | 81
units on a scale
  Week 1 | 3.66 (0.07) | 3.63 (0.07) | 3.60 (0.07) | 3.72 (0.08)
  Week 2: number analyzed (Participants) | 153 | 146 | 143 | 81
  Week 2 | 3.32 (0.08) | 3.30 (0.08) | 3.19 (0.08) | 3.26 (0.10)
  Week 3: number analyzed (Participants) | 150 | 145 | 144 | 78
  Week 3 | 3.20 (0.08) | 3.20 (0.08) | 3.14 (0.08) | 3.23 (0.10)
  Week 4: number analyzed (Participants) | 145 | 137 | 138 | 78
  Week 4 | 2.93 (0.09) | 2.93 (0.09) | 2.82 (0.09) | 2.97 (0.11)
  Week 6: number analyzed (Participants) | 143 | 136 | 136 | 78
  Week 6 | 2.70 (0.09) | 2.64 (0.10) | 2.65 (0.10) | 2.78 (0.12)
  Week 8: number analyzed (Participants) | 137 | 132 | 133 | 78
  Week 8 | 2.69 (0.10) | 2.58 (0.08) | 2.60 (0.10) | 2.57 (0.12)

10. Secondary Outcome: Percentage of Participants With CGI-S Remission
Description: CGI-S remission was defined as a CGI-S score of 1 or 2. The CGI-S provides the clinician's impression of the participant's current state of mental illness. The clinician uses his or her clinical experience of this participant population to rate the severity of the participant's current mental illness on a 7-point scale ranging from 1 (normal - not at all ill) to 7 (among the most extremely ill participants).
Time Frame: Weeks 1, 2, 3, 4, 6, and 8 of Phase B
Population: FAS included all participants randomized to the double-blind, 8-week treatment period (Phase B) who took at least 1 dose of double-blind study drug and who had a valid baseline (Week 4 of Phase A) assessment and at least 1 valid post-baseline assessment of the CDRS-R total score. Number analyzed = participants evaluable at specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind: Placebo | Double-Blind: Vortioxetine 10 mg | Double-Blind: Vortioxetine 20 mg | Double-Blind: Fluoxetine 20 mg
Number analyzed (Participants) | 153 | 148 | 148 | 81
percentage of participants
  Week 1: number analyzed (Participants) | 153 | 148 | 146 | 81
  Week 1 | 0 | 0.7 | 0 | 0
  Week 2: number analyzed (Participants) | 153 | 148 | 147 | 81
  Week 2 | 0.7 | 3.4 | 1.4 | 3.7
  Week 3 | 3.3 | 4.1 | 4.7 | 7.4
  Week 4 | 8.5 | 8.1 | 12.8 | 12.3
  Week 6 | 14.4 | 16.2 | 16.2 | 14.8
  Week 8 | 22.9 | 22.3 | 20.9 | 29.6

11. Secondary Outcome: Change From Baseline in Children's Global Assessment Scale (CGAS) Score at Weeks 4 and 8 of Phase B
Description: The CGAS is a clinician-rated global scale to measure the lowest level of functioning for a child (4 to 16 years) during a specified time period. The CGAS contains behaviourally-oriented descriptors at each anchor point that depict behaviours and life situations applicable to a child. The score ranges from 1 (most functionally impaired child) to 100 (the healthiest). A score greater than 70 indicates normal function.
Time Frame: Baseline (Week 4 of Phase A), Weeks 4 and 8 of Phase B
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-Blind: Placebo | Double-Blind: Vortioxetine 10 mg | Double-Blind: Vortioxetine 20 mg | Double-Blind: Fluoxetine 20 mg
Number analyzed (Participants) | 146 | 139 | 142 | 79
units on a scale
  Change at Week 4 | 8.93 (1.23) | 9.84 (1.25) | 8.73 (1.26) | 10.54 (1.39)
  Change at Week 8: number analyzed (Participants) | 136 | 132 | 134 | 78
  Change at Week 8 | 12.71 (1.31) | 12.98 (1.33) | 13.22 (1.34) | 16.35 (1.51)

12. Secondary Outcome: Change From Baseline in Pediatric Quality of Life Inventory (PedsQL) Visual Analogue Scales (VAS): Afraid or Scared (Anxiety) Score at Weeks 4 and 8 of Phase B
Description: The PedsQL™ VAS is designed to measure at-that-moment functioning in children and adolescents. The PedsQL VAS consists of 6 domains: anxiety, sadness, anger, worry, fatigue and pain using visual analogue scales. The functionality for each domain is measured on a 10 cm line with a happy face at one end and a sad face at the other (0-10 points). The participants are asked to mark on the line how they feel. A lower value represents a better outcome.
Time Frame: Baseline (Week 4 of Phase A), Weeks 4 and 8 of Phase B
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-Blind: Placebo | Double-Blind: Vortioxetine 10 mg | Double-Blind: Vortioxetine 20 mg | Double-Blind: Fluoxetine 20 mg
Number analyzed (Participants) | 145 | 139 | 141 | 79
units on a scale
  Change at Week 4 | -0.48 (0.27) | -0.51 (0.27) | -0.48 (0.27) | -0.41 (0.31)
  Change at Week 8: number analyzed (Participants) | 136 | 130 | 134 | 78
  Change at Week 8 | -0.73 (0.26) | -1.07 (0.27) | -1.01 (0.27) | -1.08 (0.29)

13. Secondary Outcome: Change From Baseline in PedsQL VAS: Sad or Blue (Sadness) Score at Weeks 4 and 8 of Phase B
Description: as for outcome 12
Time Frame: Baseline (Week 4 of Phase A), Weeks 4 and 8 of Phase B
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-Blind: Placebo | Double-Blind: Vortioxetine 10 mg | Double-Blind: Vortioxetine 20 mg | Double-Blind: Fluoxetine 20 mg
Number analyzed (Participants) | 145 | 139 | 141 | 79
units on a scale
  Change at Week 4 | -1.20 (0.31) | -1.65 (0.31) | -1.78 (0.31) | -1.42 (0.35)
  Change at Week 8: number analyzed (Participants) | 136 | 130 | 134 | 78
  Change at Week 8 | -1.72 (0.32) | -2.23 (0.32) | -2.05 (0.32) | -2.31 (0.36)

14. Secondary Outcome: Change From Baseline in PedsQL VAS: Angry Score at Weeks 4 and 8 of Phase B
Description: as for outcome 12
Time Frame: Baseline (Week 4 of Phase A), Weeks 4 and 8 of Phase B
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-Blind: Placebo | Double-Blind: Vortioxetine 10 mg | Double-Blind: Vortioxetine 20 mg | Double-Blind: Fluoxetine 20 mg
Number analyzed (Participants) | 144 | 139 | 140 | 79
units on a scale
  Change at Week 4 | -0.98 (0.30) | -1.36 (0.31) | -1.33 (0.31) | -1.22 (0.35)
  Change at Week 8: number analyzed (Participants) | 136 | 130 | 133 | 78
  Change at Week 8 | -1.24 (0.31) | -1.98 (0.32) | -1.36 (0.32) | -1.67 (0.36)

15. Secondary Outcome: Change From Baseline in PedsQL VAS: Worry Score at Weeks 4 and 8 of Phase B
Description: as for outcome 12
Time Frame: Baseline (Week 4 of Phase A), Weeks 4 and 8 of Phase B
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-Blind: Placebo | Double-Blind: Vortioxetine 10 mg | Double-Blind: Vortioxetine 20 mg | Double-Blind: Fluoxetine 20 mg
Number analyzed (Participants) | 145 | 139 | 141 | 79
units on a scale
  Change at Week 4 | -0.63 (0.31) | -1.48 (0.32) | -1.21 (0.32) | -1.27 (0.36)
  Change at Week 8: number analyzed (Participants) | 136 | 130 | 134 | 78
  Change at Week 8 | -1.08 (0.32) | -1.82 (0.33) | -1.45 (0.33) | -1.41 (0.36)

16. Secondary Outcome: Change From Baseline in PedsQL VAS: Tired (Fatigue) Score at Weeks 4 and 8 of Phase B
Description: as for outcome 12
Time Frame: Baseline (Week 4 of Phase A), Weeks 4 and 8 of Phase B
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-Blind: Placebo | Double-Blind: Vortioxetine 10 mg | Double-Blind: Vortioxetine 20 mg | Double-Blind: Fluoxetine 20 mg
Number analyzed (Participants) | 145 | 139 | 141 | 79
units on a scale
  Change at Week 4 | -1.22 (0.34) | -1.19 (0.35) | -1.63 (0.35) | -0.94 (0.39)
  Change at Week 8: number analyzed (Participants) | 136 | 130 | 134 | 78
  Change at Week 8 | -1.39 (0.36) | -1.32 (0.37) | -1.74 (0.37) | -1.73 (0.41)

17. Secondary Outcome: Change From Baseline in PedsQL VAS: Pain or Hurt Score at Weeks 4 and 8 of Phase B
Description: as for outcome 12
Time Frame: Baseline (Week 4 of Phase A), Weeks 4 and 8 of Phase B
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-Blind: Placebo | Double-Blind: Vortioxetine 10 mg | Double-Blind: Vortioxetine 20 mg | Double-Blind: Fluoxetine 20 mg
Number analyzed (Participants) | 145 | 139 | 141 | 79
units on a scale
  Change at Week 4 | -0.22 (0.28) | -0.81 (0.28) | -0.45 (0.28) | -0.50 (0.32)
  Change at Week 8: number analyzed (Participants) | 136 | 130 | 134 | 78
  Change at Week 8 | -0.70 (0.28) | -0.79 (0.28) | -1.02 (0.28) | -0.69 (0.32)

18. Secondary Outcome: Change From Baseline in PedsQL VAS Total Average Score at Weeks 4 and 8 of Phase B
Description: The PedsQL™ VAS is designed to measure at-that-moment functioning in children and adolescents. The PedsQL™ VAS consists of 6 domains: anxiety, sadness, anger, worry, fatigue, and pain using visual analogue scales. The functionality for each domain is measured on a 10cm line with a happy face at one end and a sad face at the other (0-10 points). The participants are asked to mark on the line how they feel. The total score is the average of all 6 items. A lower value represents a better outcome.
Time Frame: Baseline (Week 4 of Phase A), Weeks 4 and 8 of Phase B
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-Blind: Placebo | Double-Blind: Vortioxetine 10 mg | Double-Blind: Vortioxetine 20 mg | Double-Blind: Fluoxetine 20 mg
Number analyzed (Participants) | 145 | 139 | 141 | 79
units on a scale
  Change at Week 4 | -0.81 (0.19) | -1.19 (0.19) | -1.17 (0.20) | -1.01 (0.22)
  Change at Week 8: number analyzed (Participants) | 136 | 130 | 134 | 78
  Change at Week 8 | -1.17 (0.20) | -1.55 (0.20) | -1.47 (0.20) | -1.54 (0.23)

19. Secondary Outcome: Change From Baseline in PedsQL Emotional Distress Summary Average Score at Weeks 4 and 8 of Phase B
Description: The PedsQL™ VAS is designed to measure at-that-moment functioning in children and adolescents. The PedsQL VAS consists of 6 domains: anxiety, sadness, anger, worry, fatigue and pain using visual analogue scales. The functionality for each domain is measured on a 10 cm line with a happy face at one end and a sad face at the other (0-10 points). The participants are asked to mark on the line how they feel. The average emotional distress summary score is the mean of the anxiety, sadness, anger, and worry items. A lower value represents a better outcome.
Time Frame: Baseline (Week 4 of Phase A), Weeks 4 and 8 of Phase B
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-Blind: Placebo | Double-Blind: Vortioxetine 10 mg | Double-Blind: Vortioxetine 20 mg | Double-Blind: Fluoxetine 20 mg
Number analyzed (Participants) | 145 | 139 | 141 | 79
units on a scale
  Change at Week 4 | -0.84 (0.21) | -1.28 (0.21) | -1.22 (0.22) | -1.13 (0.24)
  Change at Week 8: number analyzed (Participants) | 136 | 130 | 134 | 78
  Change at Week 8 | -1.22 (0.22) | -1.80 (0.22) | -1.51 (0.22) | -1.66 (0.25)

20. Secondary Outcome: Change From Baseline in Paediatric Quality of Life Enjoyment and Satisfaction Questionnaire (PQ-LES-Q) Total Score (Items 1 to 14) at Weeks 4 and 8 of Phase B
Description: The PQ-LES-Q is a patient-rated scale designed to assess satisfaction with life. It is an adaptation of the Quality of Life Enjoyment and Satisfaction Questionnaire, which is used to measure quality of life in adults. The PQ-LES-Q consist of 15 items, item 1 to 14 assess the degree of satisfaction experienced by participants in various areas of daily functioning, and item 15 allows subjects to summarise their experience in a global rating. Each item is rated on a 5-point scale from 1 (very poor) to 5 (very good). The total score range of item 1 to 14 is 14 to 70, with higher scores indicating greater satisfaction.
Time Frame: Baseline (Week 4 of Phase A), Weeks 4 and 8 of Phase B
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-Blind: Placebo | Double-Blind: Vortioxetine 10 mg | Double-Blind: Vortioxetine 20 mg | Double-Blind: Fluoxetine 20 mg
Number analyzed (Participants) | 145 | 139 | 140 | 79
units on a scale
  Change at Week 4 | 3.94 (0.95) | 4.90 (0.96) | 4.90 (0.97) | 4.36 (1.09)
  Change at Week 8: number analyzed (Participants) | 136 | 132 | 134 | 78
  Change at Week 8 | 6.22 (0.98) | 7.08 (0.99) | 7.14 (1.00) | 6.79 (1.12)

21. Secondary Outcome: Change From Baseline in PQ-LES-Q Overall Evaluation Score (Item 15) at Weeks 4 and 8 of Phase B
Description: The PQ-LES-Q is a patient-rated scale designed to assess satisfaction with life. It is an adaptation of the Quality of Life Enjoyment and Satisfaction Questionnaire, which is used to measure quality of life in adults. The PQ-LES-Q consist of 15 items, item 1 to 14 assess the degree of satisfaction experienced by participants in various areas of daily functioning, and item 15 allows subjects to summarize their experience in a global rating. Item 15 is rated on a 5-point scale from 1 (very poor) to 5 (very good).
Time Frame: Baseline (Week 4 of Phase A), Weeks 4 and 8 of Phase B
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-Blind: Placebo | Double-Blind: Vortioxetine 10 mg | Double-Blind: Vortioxetine 20 mg | Double-Blind: Fluoxetine 20 mg
Number analyzed (Participants) | 145 | 139 | 140 | 79
units on a scale
  Change at Week 4 | 0.28 (0.09) | 0.37 (0.09) | 0.43 (0.09) | 0.24 (0.11)
  Change at Week 8: number analyzed (Participants) | 136 | 132 | 134 | 78
  Change at Week 8 | 0.41 (0.09) | 0.49 (0.09) | 0.52 (0.09) | 0.45 (0.11)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 16
Description: All-patients-treated set Phase A (APTS_A) included all participants enrolled to the 4-week Single-blind period (Phase A) who received at least 1 dose of study drug. All-patients-treated set Phase B (APTS) included all participants randomized to the double-blind, 8-week treatment period (Phase B) who took at least 1 dose of double-blind study drug.
Arm/Group | Single-Blind: Placebo | Double-Blind: Placebo | Double-Blind: Vortioxetine 10 mg | Double-Blind: Vortioxetine 20 mg | Double-Blind: Fluoxetine 20 mg
All-Cause Mortality (participants affected / at risk) | 0/677 | 0/153 | 0/151 | 0/153 | 0/83
Serious Adverse Events (participants affected / at risk) | 6/677 | 3/153 | 1/151 | 2/153 | 1/83
Other Adverse Events (participants affected / at risk) | 106/677 | 45/153 | 55/151 | 42/153 | 27/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single-Blind: Placebo (N=677) | Double-Blind: Placebo (N=153) | Double-Blind: Vortioxetine 10 mg (N=151) | Double-Blind: Vortioxetine 20 mg (N=153) | Double-Blind: Fluoxetine 20 mg (N=83)
Suicide attempt (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intentional self-injury (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Tracheitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mania (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single-Blind: Placebo (N=677) | Double-Blind: Placebo (N=153) | Double-Blind: Vortioxetine 10 mg (N=151) | Double-Blind: Vortioxetine 20 mg (N=153) | Double-Blind: Fluoxetine 20 mg (N=83)
Abdominal pain upper (Gastrointestinal disorders) | 15 (16) | 4 (4) | 4 (6) | 3 (4) | 3 (3)
Nausea (Gastrointestinal disorders) | 23 (23) | 7 (7) | 19 (22) | 17 (25) | 5 (6)
Headache (Nervous system disorders) | 39 (54) | 17 (23) | 14 (19) | 14 (16) | 4 (5)
Abdominal pain (Gastrointestinal disorders) | 9 (9) | 2 (2) | 9 (11) | 6 (8) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 9 (9) | 4 (5) | 5 (5) | 1 (1) | 3 (6)
Dry mouth (Gastrointestinal disorders) | 5 (5) | 4 (4) | 4 (4) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 13 (13) | 3 (3) | 14 (20) | 10 (16) | 3 (3)
Illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (8) | 0 (0)
Nasopharyngitis (Infections and infestations) | 13 (13) | 5 (8) | 6 (8) | 4 (4) | 3 (3)
Viral infection (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Weight increased (Investigations) | 1 (1) | 4 (4) | 1 (1) | 3 (3) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (2) | 2 (2) | 3 (4)
Dizziness (Nervous system disorders) | 9 (10) | 5 (5) | 7 (7) | 5 (5) | 3 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-08-21): https://cdn.clinicaltrials.gov/large-docs/55/NCT02709655/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-08): https://cdn.clinicaltrials.gov/large-docs/55/NCT02709655/SAP_001.pdf